CLINICAL TRIAL: NCT05008003
Title: Vit D3 Adjuvant Therapy for Early Mild Symptoms of COVID-19
Brief Title: Vit D3 for Early Symptoms of COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ayub Teaching Hospital (Other)
Collaborators: Liaquat University of Medical & Health Sciences (Other)
Responsible Party: Principal Investigator, Dr Umer Farooq, Professor of Community Medicine, Ayub Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQC/COVID/08-2021
Record Dates: First submitted 2021-08-11; First posted 2021-08-17 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): This arm will receive the standard of care as per the hospital guidelines.
  Interventions: Drug: Standard of care
- Investigational treatment (Experimental): This arm will receive vitamin D3 supplement as add-on to the standard of care.
  Interventions: Drug: Standard of care; Dietary Supplement: Vitamin D3

INTERVENTIONS:
Drug: Standard of care — Standard of care treatment as per the hospital guidelines
Dietary Supplement: Vitamin D3 — A daily dose of 5000 IU vitamin D3 for 7 days.
  Arms: Investigational treatment

SUMMARY:
This study is aimed to investigate the treatment vitamin D3 as complementary therapy with routine care for early mild symptoms of COVID-19 in outpatients setting.

DETAILED DESCRIPTION:
There is currently no specific early-stage therapeutic treatment available for COVID-19.

Vitamin D3 is a strong antioxidant, and anti-inflammatory/immunomodulatory agent.

The present study is aimed to investigate the treatment benefits of vitamin D3 as add-on therapy to the routine care for early mild symptoms of COVID-19 infection in outpatients setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older, of either gender
* Patients must be tested positive for SARS-CoV-2 by RT-PCR
* Patients must exhibit typical symptoms of COVID-19 disease at screening such as fever, fatigue, a dry and contagious cough, loss of appetite, body aches, shortness of breath, mucus or phlegm, sore throat, headache, chills, sometimes withshaking, loss of smell or taste, congestion or runny nose, nausea, or vomiting, diarrhea, muscular pain etc.
* Patients must be in the early stage of COVID-19 disease who do not require hospitalization at the time of screening
* Patients must be under the care of a Physician for diagnosis of COVID-19
* Patients who have signed informed consent

Exclusion Criteria:

* Patients with proven hypersensitivity or allergic reaction to quercetin or curcumin
* Patients with known chronic kidney disease with estimated creatinine clearance < 50 mL/minute or need for dialysis
* Patients who are severely hypotensive defined as needing hemodynamic pressors to maintain blood pressure
* Patients taking anticoagulant/antiplatelet drugs such as Coumarine, Heparine, Aspirin, Clopidrogel, dalteparin, enoxaparin, ticlopidine and warparin.
* Patients with gallstone obstruction
* Hypothyroid suppering patients
* Patients with moderate or severe thrombocytopenia (platelet count <100 ×10⁹/L);
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-02 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 Negativity by RT-PCR | From day 1 to day 14
  The numbers of patients that tests COVID-19 negative
COVID-19 symptoms improvement | From day 1 to day 14
  The numbers of patients whose COVID-19 symptoms are subsided

SECONDARY OUTCOMES:
Changes in CRP level | From day 1 to day 14
  Improvement in blood CRP level
Changes in D-dimer level | From day 1 to day 14
  Improvement in blood D-dimer level
Changes in LDH level | From day 1 to day 14
  Improvement in blood LDH level
Changes in ferritin level | From day 1 to day 14
  Improvement in blood ferritin level
Changes in full blood count | From day 1 to day 14
  Improvement in full blood count

CONTACTS AND LOCATIONS:
Locations (1):
- Ayub Teaching Hospital, Abbottabad, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No